CLINICAL TRIAL: NCT01818466
Title: Anterior Tibiotalar Arthrodesis With Blade Plate Fixation in Treatment of Post-traumatic Arthritis Secondary to Pilon Fracture
Brief Title: Anterior Tibiotalar Arthrodesis With Blade Plate Fixation
Status: Withdrawn | Type: Observational
Why Stopped: Dr. Higgins does not have a sub-investigator that can complete the study.
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Thomas Higgins, M.D., University of Utah
Other Study IDs: 57171
Record Dates: First submitted 2013-02-05; First posted 2013-03-26 (Estimated); Last update posted 2016-06-28 (Estimated); Status verified 2016-06

CONDITIONS: Pilon Fracture; Arthritis
MeSH Terms: conditions — Arthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of this study is to evaluate the clinical and radiographic outcomes of patients who have previously undergone tibiotalar arthrodesis using an anterior approach with blade-plate fixation for tibiotalar arthritis secondary to injury to the articular surface of the distal tibia.

ELIGIBILITY:
Inclusion Criteria:

* All patients whom have undergone anterior ankle arthrodesis with a blade plate construct, performed by a single surgeon, between January 2003 and July 2011 at the University of Utah or Primary Childrens Medical Center (PCMC) will be eligible for inclusion.

Exclusion Criteria:

* Any patient who is not 18 years of age or older will not be eligible for the study.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have previously undergone tibiotalar arthrodesis using an anterior approach with blade-plate fixation for tibiotalar arthritis secondary to injury to the articular surface of the distal tibia.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2012-11; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Outcome Questionnaires relating to the patients current condition | 1 Year after Surgery
  These questionnaires will include the FAOS, FADI, SF-36, PromisCAT, SMFA, and the DRAM.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Higgins, MD, Principal Investigator — Orthopedic Surgery Operations